CLINICAL TRIAL: NCT05569447
Title: Tree Branch Penetrating Injury Into Zone III of the Neck
Brief Title: Tree Branch Penetrating Injury
Status: Completed | Type: Observational
Sponsor: South Texas Health System McAllen (Other)
Responsible Party: Principal Investigator, Dr. Carlos H. Palacio, Trauma Surgeon, South Texas Health System McAllen
Other Study IDs: D-22-01107
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Penetrating Injury Neck
MeSH Terms: interventions — Balloon Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Balloon Tamponade — A tamponade device that was fashioned using an 18F red rubber catheter and Penrose drain that was cut to the approximate length of the tract and ligated proximally and distally with #0 silk.

SUMMARY:
Penetrating trauma to the neck can result in severe morbidity and mortality. Location of the injury dictates the appropriate clinical management. Challenging traumatic injuries require resourceful treatment options

DETAILED DESCRIPTION:
A complex traumatic case of a foreign body penetrating the neck, the parotid gland, disrupting the internal jugular vein, with the tip resting at the anterior aspect of the C1 ring is reported. In this case, the authors seek to describe the clinical management of a vascular injury that resulted from penetrating zone III of the neck.

Due to the complex and dense presence of various structure in the neck, injuries can be difficult to manage. Thus, an algorithm identifies management strategies that are suggested based on the location of the injury, signs of vascular injury, identified injured structures and the hemodynamic stability of the patient. Balloon tamponade has been described in other organs of the body and it might be a therapeuticn option in patients were venous injuries are difficult to access.

Penetrating neck injuries continue to result in significant morbidity and mortality. However, with appropriate and efficient evaluation and management, better outcomes are expected as demonstrated in this case.

ELIGIBILITY:
Inclusion Criteria:

* Penetrating Injury to the Neck

Exclusion Criteria:

* N?A

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma penetrating injury to the neck
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- STHS McAllen, McAllen, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided